CLINICAL TRIAL: NCT05729828
Title: Psychometric Properties of the SMART Feeding Tool
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 21.001E
Record Dates: First submitted 2023-01-23; First posted 2023-02-15 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Feeding; Difficult, Newborn; Premature Infant Disease; Dysphagia of Newborn; Nurse's Role; Feeding Disorder of Infancy or Early Childhood; Trauma and Stressor Related Disorders; Deglutition Disorders in Infants; Malnutrition, Infant
Keywords: neonate; dysphagia; trauma informed care; infant and family centred developmental care; synactive developmental theory; psychometrics; deglutition; pediatric feeding disorder; SMART Tool; life course health development
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Infant Nutrition Disorders; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: Neonates with PMA 33 weeks, 0 days or more, present in NICU. No intervention was done.

SUMMARY:
This observational study aims to evaluate the psychometric properties of a new infant feeding tool called "SMART Tool" in the neonatal intensive care unit. The main questions it aims to answer are:

1. To design a feeding tool to assess oral motor and neurobehavioral skills in neonates
2. To establish psychometrics of the new tool by doing reliability and validity tests.

DETAILED DESCRIPTION:
Research supports the use of infant-directed feeding practices versus a volume-driven approach. Infant-directed feeding practices provide developmentally supportive and neuroprotective care to fragile feeders. In addition, various assessment tools exist to evaluate both breast and bottle feeding. Assessment tools are crucial to feeders with guidance in their decision-making, identifying when an infant is ready to feed and recognizing any feeding-related safety concerns.

The scoring of a tool should provide an opportunity to reflect on the strengths and areas of deficit in feeding events and allow feeders to modify feeding practices for the next attempt or pursue further assessment by a feeding specialist. Few tools exist to evaluate both oral skills and neurobehavioral skills. Some tools available have inadequate psychometric data to support their use. If robust psychometrics exist, the length and complexity of the device may intimidate users and deter consistent use.

The SMART tool was developed to capture the multifaceted aspects of feeding while remaining brief in its administration time. The tool provides an opportunity to evaluate skills and develop a plan after feeding to provide consistent quality care. Additionally, tracking scores over time helps in patient safety for the goal of a high-reliability organization.

This study has two objectives: 1. to create a new tool using synactive development theory and trauma-informed care approach for neonates and 2. to establish this tool's psychometrics (validity and reliability). This multicenter trial will be done over four sites (NICU) in Advocate Aurora Health (AAH) to observe feeding events in neonates. Before and after each feed, scoring of feeding quality will be done to do psychometrics. If the study succeeds, this tool will be employed in clinical care in all the NICUs of AAH.

Acronyms & Abbreviations:

* AAH: Advocate Aurora Health
* NEOA: Neonatal Eating Outcome Assessment Tool
* NICU: Neonatal Intensive care unit
* PMA: Postmenstrual age (weeks)
* SMART: State of Arousal, Motor Tone, Autonomic Instability, Response to Stimulation, Total Oral Skills

ELIGIBILITY:
Inclusion Criteria:

1. At least 33 weeks, 0 days PMA
2. Able to tolerate enteral feedings
3. Parental consent available

Exclusion Criteria:

1) Respiratory support of more than two liter-per-minute oxygen via nasal cannula

Ages: 33 Weeks to 50 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates above 33 weeks, 0 days PMA in NICU
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Criteria Validity: Compare SMART Tool vs. NEOA Tool (version 5.8) Scores | 12 months
  The scale of the two tools is as follows: NEOA: feeding challenge (18 to 57), questionable (58 to 76), normal (77 to 90). SMART: caution (under 60), developing (60 to 90), capable (above 90). Higher scores are better on both scales.
  Sample size = 50 feeding events. Observers will not do any intervention. Data analysis: post-feed scores per feeding event.
Inter Rater Reliability of SMART Tool | 12 months
  Using SMART Tool, two observers will rate one feeding event of an infant. Observers = 2, Feedings events = 10. Observers will not do any intervention. Data analysis: pre-feed and post-feed scores per feeding event.
Test Retest Reliability of SMART Tool | 12 months
  Using SMART Tool, one observer will rate two feeding events of the same infant. Observer = 1, Feedings events = 20 The observer will not do any intervention. Data analysis: pre-feed and post-feed scores per feeding event.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Mishra, MD, FAAP, Principal Investigator — Advocate Health; Anne Albi, SLP, IBCLC, Principal Investigator — Advocate Health; Cynthia Liracrame, MSN, RNC-NIC, Principal Investigator — Advocate Health
Locations (4):
- United States (4):
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Advocate Children's Hospital - Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital - Park Ridge, Park Ridge, Illinois

IPD SHARING:
Plan to Share IPD: No
Not sharing